CLINICAL TRIAL: NCT00492700
Title: A One-Year, Randomized, Double-Blind, Placebo-Controlled Trial of Rosiglitazone in Non-Alcoholic Steatohepatitis
Acronym: FLIRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association pour la Recherche sur les Maladies Hépatiques Virales (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIDO-Trials-01
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2007-06

CONDITIONS: Non Alcoholic Steatohepatitis
Keywords: steatosis,; fibrosis,; diabetes,; obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Fibrosis; Diabetes Mellitus; Obesity | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
This study is intended to find out whether treatment with rosiglitazone improves the state of the liver and related blood markers in patients with nonalcoholic steatohepatitis (NASH).

DETAILED DESCRIPTION:
Phase one : A double blind randomized placebo controlled trial of rosiglitazone

* 64 pts with biopsy proven NASH will be randomized to receive either rosiglitazone 8 mg/day or placebo for one year.
* after one year of treatment patients will undergo a liver biopsy then a 4 month follow off treatment

Primary endpoint: improvement of at least 30% of the histological score of steatosis Secondary endpoints: improvement in ALT values, in necrosis and inflammation and fibrosis

Phase II extension open label trial

All participants to the phase one regardless of the drug received in the first year will be treated with rosiglitazone for 2 additional years. A liver biopsy will be performed at the end of these two additional years in order to find out whether prolonged rosiglitazone therapy further results in improvement of liver injury in NASH patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NASH with steatosis >= 20%
* Increased serum ALT

Exclusion Criteria:

* bland steatosis
* daily alcohol > 20/30 g (women/men)
* any other cause of liver disease
* secondary NASH including drug-induced steatohepatitis
* treatment with insulin or glitazones
* cardiac insufficiency
* Hb < 10 g/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-01

PRIMARY OUTCOMES:
improvement in steatosis

SECONDARY OUTCOMES:
improvement in transaminase levels; improvement/less worsening in necrosis and inflammatory activity and /or fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Ratziu, MD PhD, Principal Investigator — Hôpital Pitié Salpêtrière, APHP
Locations (1):
- Service d'hépatogastroenérologie, Hôpital Pitié Salpêtrière, Paris, France

REFERENCES:
- [Derived] Ratziu V, Charlotte F, Bernhardt C, Giral P, Halbron M, Lenaour G, Hartmann-Heurtier A, Bruckert E, Poynard T; LIDO Study Group. Long-term efficacy of rosiglitazone in nonalcoholic steatohepatitis: results of the fatty liver improvement by rosiglitazone therapy (FLIRT 2) extension trial. Hepatology. 2010 Feb;51(2):445-53. doi: 10.1002/hep.23270. PMID 19877169